CLINICAL TRIAL: NCT01644071
Title: Genetic-pharmacological Neuroimaging of the Serotonergic System in Violent Video Games
Brief Title: Serotonergic System and Violent Video Games
Acronym: Serogen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: CTC-A_12-023
Record Dates: First submitted 2012-06-20; First posted 2012-07-18 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Healthy Volunteers
Keywords: violent video games; serotonergic system
MeSH Terms: interventions — Dexetimide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- arm 1 (Experimental): application of three treatments and three masurements within 3 weeks
  Interventions: Drug: cipralex

INTERVENTIONS:
Drug: cipralex — one time 10 mg, tablet

SUMMARY:
Aggressive behavior (AB) is a major burden to society with severe socio-economic consequences. Genetic studies suggest a high heritability of AB; in particular, the low expressing allele of the MAOA gene (MAOA-L) has been associated with increased AB. Recent neural aggression models have suggested a dysfunctional emotion regulation circuit including amygdala, orbitofrontal, and anterior cingulate cortex. Dysregulated serotonergic (5-HT) projections from the anterior cingulate cortex to the amygdala have been suggested to promote aggressive behavior. This finding is well in line with the observation that the MAOA-L allele leads to a reduced expression of monoamine oxidase A and thus to an overflow of 5-HT in serotonergic cortico-amygdalar projections. However, due to methodological and ethical constraints, the neural substrates of AB are difficult to assess. A possible solution is the use of virtual violence which permits AB against virtual characters without direct consequences for any real person and can be easily applied in functional imaging experiments. There is evidence that virtual and real aggression share common neural substrates. AB in violent video games inhibits rostral anterior cingulate cortex (ACC) and amygdala in line with the suggested neurophysiological circuits underlying real-life AB.

DETAILED DESCRIPTION:
Our study plan comprises the assessment of brain activation patterns during virtual AB in a violent video game with functional magnetic resonance imaging under three experimental conditions in randomized, double-blind fashion:

1. Increase of synaptic 5-HT with a selective serotonin reuptake inhibitor (SSRI, Cipralex ®);
2. reduction of synaptic 5-HT with the Rapid Tryptophan Depletion Test (RTD); and 3) Placebo.

A blood sample genotyping will assess the allelic expression of the MAOA gene. We hypothesize

1. a modification of the ACC-amygdala system by the serotonergic intervention and
2. an interaction with the genotype concerning the MAOA gene. The results of this study will give valuable insights into the neurogenetic biology underlying aggression which will open new perspectives for therapeutical and pharmacological intervention.

ELIGIBILITY:
Inclusion Criteria:

* male
* age 18-60 (adults), age 12-17 (juveniles)
* right-handedness
* German native language

Exclusion Criteria:

* any contraindications against MR investigations
* any contraindications against application of SSRIs
* any history of neurological or psychiatric illness
* history of drug abuse
* history of psychopharmacological therapy

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2012-02; Primary Completion 2014-02 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
functional neuroimaging | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, Psychotherapy and Psychosomatics, University Hospital Aachen, Aachen, Germany